CLINICAL TRIAL: NCT04357301
Title: Tight Systolic Arterial Pressure Control Using a Closed-loop System for Vasopressor Infusion in Patients Undergoing High-risk Abdominal Surgery: A Proof-of-Concept Study
Brief Title: Tight Closed-loop Systolic Arterial Pressure Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Alexandre Joosten, MD PhD, Principal Investigator, Erasme University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P2020/157
Record Dates: First submitted 2020-04-19; First posted 2020-04-22 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Single prospective pilot study (12 patients)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Closed-loop (Experimental): Closed-loop administration of norepinephrine
  Interventions: Device: Closed-loop vasopressor

INTERVENTIONS:
Device: Closed-loop vasopressor — The system will adjust the norepineprhine infusion rate based on a target SAP of 130 mmHg in 20 patients

SUMMARY:
The purpose of this case series is to evaluate the performance of a novel closed-loop (automated) vasopressor administration system that delivers norepinephrine using feedback from standard operating room hemodynamic monitoring (EV1000 monitoring device, Edwards Lifesciences, Irvine, USA).

DETAILED DESCRIPTION:
In this case series, the investigators will report the percentage of case time in hypotension (defined as systolic arterial pressure (SAP) < 117mmHg). The target mean arterial pressure (MAP) will be set at a SAP of 130mmHg in all patients. Definition of Hypotension is target SAP - 10% (130mmHg - 13 mmHg = 117 mmHg). We will use the same SAP target in all patients even if we used a modified definition of hypotension from the study of Futier and colleagues ( JAMA 2017). We won't use a individualized SAP for each patient but the same SAP target in all patients.

The investigators want to demonstrate that the closed-loop system can prevent hypotension at this specific set point.

The Investigators have shown the system works well based on a target MAP but not yet using a target of SAP.

The investigators will test the system in a pilot study of 13 patients undergoing High-risk abdominal surgery which require the placement of a arterial catheter, the optimization of fluid therapy and a tight SAP control.

Participants will receive standard patient care in that in no way will their anesthetic or surgical procedure will be altered as part of the study, with the exception of vasopressor administration ( automatically delivery instead of manually adjustments)

Fluids will be given as goal directed fluid therapy in order to maintain stroke volume variation below 13% (hospital guidelines).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age of >17)
* Elective high-risk abdominal surgery
* Patients with an arterial line and in whom a goal directed fluid therapy protocol is applied manually (administration of fluid bolus to maintain a stroke volume variation < 13%)

Exclusion Criteria:

* Atrial Fibrillation
* Pregnancy
* Subjects without the capacity to give informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Percentage of case Time in hypotension (SAP <117 mmHg) | At postoperative day 1
  The primary outcome will be the percentage of case time in predefined SAP target (SAP of 130 mmHg -10 % = 117 mmHg)

SECONDARY OUTCOMES:
Amount of vasopressors received | At postoperative day 1
  Amount of vasopressors received (norepinephrine)
Number of vasopressors infusion rate modifications | At postoperative day 1
  Number of vasopressors infusion rate modifications
Percentage of case time with a MAP < 65 mmHg | At postoperative day 1
  Percentage of case time with a MAP < 65 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Joosten, MD PhD, Principal Investigator — ERASME
Locations (1):
- Erasme, Brussels, Belgium